CLINICAL TRIAL: NCT01139307
Title: Development of Novel Therapeutics for AMKL
Brief Title: Biomarkers in Samples From Patients With Down Syndrome and Acute Megakaryoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B1; COG-AAML10B1 (Other: Children's Oncology Group); CDR0000671427 (Other: Clinical Trials.gov); NCI-2011-02218 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-05; First posted 2010-06-08 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia
Keywords: adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute | interventions — Cell Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cell culture procedure
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood or tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in samples from patients with Down syndrome and acute megakaryoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether megakaryocyte differentiation agents comprising a Rho kinase inhibitor and a JAK3 inhibitor can lead to proliferation arrest, polyploidization, and terminal differentiation of blasts in specimens from patients with Down syndrome and acute megakaryoblastic leukemia.

OUTLINE: Cryopreserved specimens are cultured and treated in vivo (in mice) and in vitro with megakaryocytic differentiation agents comprising a Rho kinase inhibitor and a JAK3 inhibitor.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute megakaryoblastic leukemia
* Diagnosis of Down syndrome
* Cryopreserved specimens available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of acute megakaryoblastic leukemia or diagnosis of Down syndrome when cryopreserved specimens are available.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proliferation arrest
Polyploidization
Terminal differentiation

CONTACTS AND LOCATIONS:
Overall Officials: John Crispino, PhD, Principal Investigator — Robert H. Lurie Cancer Center